CLINICAL TRIAL: NCT03967327
Title: A Study to Evaluate the Efficacy and Safety of Buprenorphine Transdermal Patch Compared to Morphine Sulfate Sustained-release Tablet in Opioid Pre-treated Chinese Subjects With Moderate to Severe Chronic Cancer Pain
Brief Title: A Study to Evaluate Buprenorphine Transdermal Patch in Chinese Subjects With Moderate to Severe Chronic Cancer Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUP14-CN-301
Record Dates: First submitted 2019-05-15; First posted 2019-05-30 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOR SR (Active Comparator): This arm includes MOR SR and placebo for BUP TDS, detailed information is as below:
  Treatment dosage form dosage frequency duration MOR SR Tablet 10,30,60mg q12h 8 weeks
  Placebo for Patch -- every 3-4 days 8 weeks BUP TDS
  Interventions: Drug: Buprenorphine transdermal patches; Drug: Morphine Sulfate Sustained-Release Tablet
- BUP TDS (Experimental): This arm includes BUP TDS and placebo for MOR SR, detailed information is as below:
  Treatment dosage form dosage frequency duration Placebo for Tablet -- q12h 8 weeks MOR SR
  BUP TDS Patch 20/30/40mg every 3-4 days 8 weeks
  Interventions: Drug: Buprenorphine transdermal patches; Drug: Morphine Sulfate Sustained-Release Tablet

INTERVENTIONS:
Drug: Buprenorphine transdermal patches — It should be applied to non-irritated, intact skin of the upper outer arm, upper chest, upper back or the side of the chest. The skin should be relatively hairless. If none are available, the hair at the site should be clipped, not shaven.
Drug: Morphine Sulfate Sustained-Release Tablet — It will be administered orally twice (q12h) daily.

SUMMARY:
This is a randomised, active-controlled, double-blind, double-dummy, parallel group study with BUP TDS 20 mg (release rate 35 µg/h), 30 mg (release rate 52.5 µg/h) and 40 mg (release rate 70 µg/h), and MOR SR 60 mg, 100 mg or 120 mg per day.

The study consists of 3 phases: a Pre-randomisation Phase, a Double-blind Phase and a Safety Follow-up Phase.

There will be 194 subjects to be randomized, with 97 randomized subjects in each arm to ensure 154 evaluable (per protocol population) subjects in the study.

DETAILED DESCRIPTION:
AE data are obtained by the Investigators through observation of the Subject (including examinations and investigations), from any information volunteered by the Subject and through active questioning. At each visit after informed consent has been signed, Subjects will be asked about AEs that occurred since the last visit by questioning them with regard to their well-being by "non-leading" questions. This includes AEs occurring during the administration of IMP, as well as changes in concomitant diseases (e.g. ongoing medical history). The general type of questions could be similar to "Do you have any health problems?" or "Have you had any health problems since your last clinic visit?" During blinded studies, the Subject and all personnel involved with the conduct and interpretation of the study, including the Investigators, site personnel, and the Sponsor's staff, those involved in processing and regulatory reporting of SUSARs, will be blinded to the treatment codes until unblinding. The randomisation schedule will be filed securely by the Sponsor/IRS provider in a manner such that blinding is properly maintained throughout the study. Treatment codes will not be available until unblinding, after completion of the study and data base lock, except in the case of emergency.

Statistical analyses will be performed by a designated CRO. All statistical analyses will be performed using SAS and/or other statistical software as required.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female cancer subjects, 18 years of age or older.
2. Females less than one year post-menopausal must have a negative serum pregnancy test recorded at the screening visit, be non-lactating, and willing to use adequate and reliable contraception throughout the study. Highly effective (adequate and reliable) methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilization, implants, injectables, combined oral contraceptives, some IUDs (intrauterine Device, hormonal), sexual abstinence or vasectomised partner.
3. Documented history of moderate to severe, chronic cancer pain that in the investigators' opinion requires around-the-clock opioid therapy in opioid pre-treated subjects and are likely to benefit from chronic opioid therapy through the administration of BUP TDS (20 mg, 30 mg or 40 mg) or MOR SR (60 mg/d, 100 mg/d or 120 mg/d) for the duration of the study. Subjects must be willing to discontinue their routine current opioid analgesic.
4. Subjects with inadequate therapeutic effect (inadequate analgesia or tolerability) with previous WHO step II opioids (weak opioids, e.g. tramadol, codeine) or WHO step III opioids (strong opioid) in the range of morphine equivalent dose level of 40 - 100 mg/d.

   • Moderate to severe inadequate pain at Screening visit (average pain over the last 24 hours ≥ 4 on the 0-10 NRS)
5. Estimated life expectancy ≥ 3 months.
6. Eastern Co-operative Group (ECOG) performance status of 0 - 2.
7. The antineoplastic therapies are not planned to be changed or added during the study.
8. Subjects willing and able to participate in all aspects for the study, including use of transdermal and oral medication, completion of subjective evaluations, attending scheduled clinic visits, completing telephone contacts, understanding and completing subject diary, and compliance with protocol requirements as evidenced by providing written informed consent.
9. In the investigators' opinion the subject's pre-study, non-opioid analgesics, and all other concomitant medications, including those medications for the treatment of depression, will remain stable throughout the double-blind phase of the study, and will be continued under the supervision of the investigator.
10. Subjects, who are able to read, understand and sign written informed consent prior to study participation and are willing to follow the protocol requirements.

Exclusion Criteria:

1. Any history of hypersensitivity to buprenorphine, morphine, related products, other opioids and other ingredients.
2. Subjects who have not received any opioids treatment, including WHO step II and step III opioids, for the treatment of cancer pain.
3. Subjects receiving WHO step III opioids with more than 100 mg morphine-equivalent dose per day within the last 8 weeks before the screening visit.
4. Subjects with any situation in which opioids are contra-indicated, severe respiratory depression with hypoxia and/or hypercapnia, severe chronic obstructive pulmonary disease, cor pulmonale, severe bronchial asthma, paralytic ileus, elevated carbon dioxide in the blood.
5. Evidence of clinically significant cardiovascular, renal, hepatic, or psychiatric disease, as determined by medical history, clinical laboratory tests, Electrocardiogram (ECG) results, and physical examination, that will place the subject at risk upon exposure to the study treatment or that could confound the analysis and/or interpretation of the study results.
6. Abnormal aspartate aminotransferase (AST; SGOT), alanine aminotransferase (ALT; SGPT), gamma-glutamyl transferase (GGT) or alkaline phosphatase levels (> 3 times the upper limit of normal) or an abnormal total bilirubin and/or creatinine level(s) (> 1.5 times the upper limit of normal), due to moderate to severe hepatic impairment and/or renal impairment, in the investigators' opinion.
7. Radiotherapy that, in the investigators' opinion, would influence pain during the study.
8. Cyclic chemotherapy in the 2 weeks before the screening visit or planned during the study that has shown in the past to significantly influence pain assessment or safety profile of subjects (e.g. nausea, vomiting, diarrhoea). If subjects are having their first cycle of chemotherapy during the 2 weeks before the screening visit or during the study they should be excluded.
9. Subjects with known or suspected unstable brain metastases or spinal cord compression that may require changes in systemic steroid treatment throughout the duration of the study.
10. Subjects with uncontrolled seizures.
11. Subjects with head injury, other intracranial lesions or a pre-existing increase in intracranial pressure.
12. In the investigators' opinion, subjects who are receiving antihistamines, antipsychotics, anti-anxiety agents, hypnotics, phenothiazine or other central nervous system (CNS) depressants that may pose a risk of additional CNS depression with opioid study treatments.
13. Subjects with myxoedema, not adequately treated hypothyroidism or Addison's disease.
14. Surgery completed 2 months prior to the screening visit, or planned surgery during the study that may have influence on pain during the study or preclude completion of the study.
15. Subjects receiving opioid substitution therapy for opioid addiction (e.g. methadone or buprenorphine).
16. Subjects with active alcohol or drug abuse and/or history of opioid abuse.
17. Subjects who participated in a clinical research study involving a new chemical entity or an experimental drug within 30 days of study entry (defined as the start of the Screening Period). Concurrent enrolment in another clinical trial is not permitted unless the sole purpose of the other trial at the time of the screening period is for collection of long-term follow-up/survival data.
18. Subjects taking MAO-inhibitors within 14 days prior to screening visit or throughout the study.
19. Subjects with any potential dermatological disorder at a patch application site, e.g. previous and/or current unhealed extensive dermal damage in the area where the patch was to be applied (e.g. dermatitis, burns, scarring of the skin).
20. Subjects who could not discontinue therapy that involved direct heat sources (e.g. heat lamps, electric blankets, heating pads or heated water beds) for the duration of the study.
21. Subjects with hairy areas who could not, or would not, cut the hair at the patch site for proper placement of the patch.

Additional Inclusion Criteria for Entry to Double-blind Phase:

1. Subjects continue to satisfy inclusion criteria.
2. Subject's daily MOR SR dose must be 60, 100 or 120 mg/d.
3. The MOR SR dose has been stable for at least one week prior to randomisation.
4. Subjects have achieved pain control for each day of the week before randomisation, except occasionally (no more than 3 days within the week) pain not controlled due to accidental activities or events.
5. Subjects must rate their pain (average pain over the last 24 hours based on PIS) as ≤ 3 on a 0-10 NRS with ≤ 2 doses of rescue medication for the day prior to randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-12-20 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory - Short Form (BPI-SF) | From visit 3 to study completion, as assessed up to 8 weeks
  * To demonstrate the therapeutic non-inferiority of buprenorphine transdermal patches (BUP TDS) compared to morphine sulfate sustained-release tablets (MOR SR) for the management of chronic cancer pain as assessed by the average pain over the last 24 hours on the numeric rating scale (NRS, 0-10) using the Brief Pain Inventory - Short Form (BPI-SF) (Cleeland & Ryan, 1994)
  * Moderate to severe inadequate pain at Screening visit (average pain over the last 24 hours ≥ 4 on the 0-10 NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Shukui Qin, Principal Investigator — The 81st hospital of the people's liberation army
Locations (1):
- The 81st hospital of the people's liberation army, Nanjing, China

IPD SHARING:
Plan to Share IPD: No